CLINICAL TRIAL: NCT02489097
Title: Evaluating the Incidence and Association Between Nitrous Oxide and Postoperative Cognitive Disorders in Anaesthesia
Brief Title: International Substudy Enigma2 on Postoperative Cognitive Disorders
Acronym: ISEP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis results showed futility
Sponsor: University Hospital, Geneva (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other); Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Guy Haller, Staff Anaesthetist, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAC 08-021; Enigma II nested NCT00430989 (Other: ClinicalTrials.gov)
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Anesthesia; Delirium, Dementia, Amnestic, Cognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders | interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitrous Oxide (Active Comparator): Receives a mixture of 70% Nitrous Oxide in 30% Oxygen
  Interventions: Drug: Nitrous Oxide
- Air/Oxygen (placebo) (Placebo Comparator): Receives a mixture of 70% Air in 30% Oxygen
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nitrous Oxide — Administration of a concentration of 70% Nitrous Oxide with 30% Oxygen in the anaesthetic gas mixture
  Other Names: N2O
  Arms: Nitrous Oxide
Other: Placebo — Administration of a concentration of 70% Air with 30% Oxygen in the anaesthetic gas mixture
  Other Names: Air/Oxygen
  Arms: Air/Oxygen (placebo)

SUMMARY:
The study is a substudy of the Enigma2 trial (NCT00430989) which aims at investigating the effectiveness and safety of nitrous oxide (N2O) in anaesthesia.The substudy focus is on postoperative cognitive disorders.

Substudy Hypothesis: In patients undergoing anaesthesia for major surgery, administration of N2O will reduce postoperative cognitive disorders when compared with otherwise identically managed surgical patients not receiving N2O as a component of their anaesthesia.

DETAILED DESCRIPTION:
Numerous studies questioned the routine use of nitrous oxide (N2O), the oldest anaesthetic agent used since the development of anaesthesia care. Despite its wide use, there is sufficient doubt as to the risk-benefit profile.

There is strong evidence that N2O is a major risk factor for postoperative nausea and vomiting. It is clear that (even) brief exposure to N2O impairs methionine synthetase, an enzyme required for DNA production, red and white blood cell formation. Tissue hypoxia may be more common. These adverse effects are enhanced in "sick" patients (ie. those at highest risk, with increased hospital length of stay and healthcare expenditure), and will be more likely in longer surgery. At the same time, observational studies and subgroup analysis of published trials suggest that N2O may have beneficial effects in preventing pain and postoperative cognitive disorders

Outcome trial data on postoperative cognitive disorders are lacking in this area for an anaesthetic gas used in more than 90% of all surgery around the world. The enigma2 substudy as a nested study of the large Enigma2 randomised controlled trial aims at answering this question.

The investigators aim at recruiting 420 patients in 2 of the 25 centres participating to the Enigma 2 trials, who are undergoing major surgery.

ELIGIBILITY:
Inclusion Criteria:

Adult males and females aged ≥ 45 years, undergoing noncardiac surgery and general anaesthesia that exceeds two hours.

At increased risk of cardiac events, defined as any of:

* history of coronary artery disease (angina, MI, Coronary revascularisation-Coronary Artery Bypass Graft (CABG) and Percutaneous Transluminal Coronary Angiography ( PTCA)-, positive stress testing, angiography/other imaging, Q waves on ECG)
* heart failure
* cerebrovascular disease due to atherothrombotic disease
* aortic or peripheral vascular disease

OR

three or more of the following risk factors: age ≥70 years, history of heart failure, diabetes (medicated), hypertension (medicated), preoperative serum creatinine >175 mmol/L, cholesterol ≥6.2 mmol/L, history of a transient ischemic attack (TIA),

Exclusion Criteria:

1. Dementia (MMS test≤24)
2. Parkinson Disease
3. Patients taking regularly (>2 weeks) tricyclic antidepressants or neuroleptics
4. Patients suffering from Alcohol Dependency (WHO CRITERIA )
5. Patients suffering from severe hypoacusis or visual loss or any other reason hindering the CANTAB battery testing process
6. Patients with untreated deficit in Vitamin B6, B12 and folic acid
7. Patients with marked impairment of gas-exchange requiring Fi02> 0.5 intraoperatively
8. Patients with specific circumstances where N2O is contraindicated (eg. volvulus, pulmonary hypertension, raised intracranial pressure) or the use of supplemental oxygen is planned (eg. colorectal surgery)
9. N2O unavailable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Memory, Executive function, Attention and psychomotor speed testing battery | Baseline before surgery
  Validated Computerized testing battery developed by the University of Cambridge for cognitive testing (CANTAB). Patients are tested for baseline cognitive function before surgery
Memory, Executive function, Attention and psychomotor speed using CANTAB Cognitive testing battery at 7days following surgery | First assessment (7 days)
  Validated Computerized testing battery developed by the University of Cambridge for cognitive testing (CANTAB). Patients are tested for changes from the baseline cognitive function (before surgery) at 7 days after surgery
Memory, Executive function, Attention and psychomotor speed using CANTAB Cognitive testing battery at 3 months following surgery | Second assessment (3 months)
  Validated Computerized testing battery developed by the University of Cambridge for cognitive testing (CANTAB). Patients are tested for changes from the baseline cognitive function (before surgery) at 3 months after surgery

SECONDARY OUTCOMES:
ICU stay | up to a maximum of 3 months
  Planned and unplanned admission to the ICU and ICU duration of stay; Follow up to be performed for the whole duration of hospital stay and up to a maximum of 3 months
Hospital stay | up to a maximum of 3 months
  Duration of stay in Hospital; Follow up to be performed for the whole duration of hospital stay and up to a maximum of 3 months
Quality of life | 3 months
  Use of the validated EuroQol test (EQ-5D questionnaire http://www.euroqol.org/)

CONTACTS AND LOCATIONS:
Overall Officials: Myles Paul, MD, FANZCA, Study Chair — Bayside Health
Locations (2):
- The Chinese University of Hong Kong Prince of Wales Hospital, Hong Kong, Hong Kong, China
- Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Result] Chan MTV, Wan ACM, Gin T, Leslie K, Myles PS. Chronic postsurgical pain after nitrous oxide anesthesia. Pain. 2011 Nov;152(11):2514-2520. doi: 10.1016/j.pain.2011.07.015. Epub 2011 Sep 1. PMID 21889262
- [Result] Sanders RD, Weimann J, Maze M. Biologic effects of nitrous oxide: a mechanistic and toxicologic review. Anesthesiology. 2008 Oct;109(4):707-22. doi: 10.1097/ALN.0b013e3181870a17. PMID 18813051
- [Result] Myles PS, Leslie K, Chan MT, Forbes A, Paech MJ, Peyton P, Silbert BS, Pascoe E; ENIGMA Trial Group. Avoidance of nitrous oxide for patients undergoing major surgery: a randomized controlled trial. Anesthesiology. 2007 Aug;107(2):221-31. doi: 10.1097/01.anes.0000270723.30772.da. PMID 17667565